CLINICAL TRIAL: NCT05650073
Title: Impact of Immersive Soundscapes in Outpatient Procedure Rooms on Patient Wellbeing
Brief Title: A Study of Soundscapes for Patient Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ellen C. Meltzer, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-008617
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immersive Soundscapes Environment (Experimental): Subjects having venous ablation OR port removal with Vascular Surgery at Mayo Clinic will have relaxing music and relaxing sounds played during the procedure.
  Interventions: Other: Immersive soundscapes
- Control Environment (No Intervention): Subjects having venous ablation OR port removal with Vascular Surgery at Mayo Clinic will have no music played during the procedure.

INTERVENTIONS:
Other: Immersive soundscapes — Audio technology used to create a three-dimensional sound experience in which the user is immersed in a virtual soundscape
  Arms: Immersive Soundscapes Environment

SUMMARY:
The purpose of this study is to assess the impact of immersive soundscape on patient pain, stress, anxiety, heart rate and blood pressure during an outpatient vascular surgery procedure.

DETAILED DESCRIPTION:
Adult (≥18-years-old) patients having outpatient vascular surgery procedures who elect to participate in the study will be randomized to Control/ Intervention. For Control Subjects: procedure will be performed in the procedure room with no immersive soundscape. For Intervention Subjects procedure will be performed in the procedure room with immersive soundscape.

ELIGIBILITY:
Inclusion Criteria:

- English-speaking adults

Exclusion Criteria:

* Patients needing an English interpreter
* Patients who lack the capacity to provide consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Change in Self-Report Visual Analog Pain Score | Baseline, before procedure commences, after injection of anesthetic, and end of procedure, approximately 1 hour
  Using a ruler, patients select a pain score from 0, "no pain" to 100 "intolerable pain", with a higher score indicating greater pain. The distance between "0/ no pain" and the mark indicates the pain level. The following cut points for quantifying pain using a VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Change in Self-Report Visual Analog Anxiety Score | Baseline, before procedure commences, after injection of anesthetic, and end of procedure, approximately 1 hour
  Using a ruler, patients select an anxiety score from 0, "no anxiety" to 100 "maximum anxiety imaginable", with a higher score indicating greater anxiety. The distance between "0/ no anxiety" and the mark indicates the anxiety level. Visual analogue scale for anxiety (VAS-A) has demonstrated to be a useful tool for measuring preoperative anxiety with a threshold for a clinically relevant level of anxiety at around 50mm.
Change in Self-Report Visual Analog Stress Score | Baseline, before procedure commences, after injection of anesthetic, and end of procedure, approximately 1 hour
  Using a ruler, patients select an anxiety score from 0, "no stress" to 100 "maximum anxiety imaginable", with a higher score indicating greater anxiety. The distance between "0/ no anxiety" and the mark indicates the anxiety level. Visual analogue scale for anxiety (VAS-A) has demonstrated to be a useful tool for measuring preoperative anxiety with a threshold for a clinically relevant level of anxiety at around 50mm.
Change in Heart Rate | Baseline, before procedure commences, after injection of anesthetic, and end of procedure, approximately 1 hour
  Number of beats per minute
Change in Blood Pressure | Baseline, before procedure commences, after injection of anesthetic, and end of procedure, approximately 1 hour
  Measured in millimeters of mercury (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Meltzer, MD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayoclinic.org